CLINICAL TRIAL: NCT02012920
Title: A Phase 1/2 Open-Label Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Seviteronel in Subjects With Castration-Resistant Prostate Cancer
Brief Title: A Study to Evaluate Oral VT-464 in Patients With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocrin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INO-VT-464-CL-001; VMT-VT-464-CL-001 (Other: Innocrin)
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Castration-resistant Prostate Cancer; CRPC
Keywords: castration-resistant prostate cancer; CYP17; P450c17a; lyase; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Failure of Abiraterone or Enzalutamide (Experimental): Seviteronel: given orally once daily in 28 day cycles
  Interventions: Drug: Seviteronel: given orally once daily in 28 day cycles
- Double Failure of Abiraterone and Enzalutimide (Experimental): Seviteronel: given orally once daily in 28 day cycles
  Interventions: Drug: Seviteronel: given orally once daily in 28 day cycles

INTERVENTIONS:
Drug: Seviteronel: given orally once daily in 28 day cycles

SUMMARY:
The goal of this clinical study is to determine the safety, tolerability, pharmacokinetics and activity of Seviteronel, a lyase-selective inhibitor of CYP17, in patients with castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a Phase 1/2 study of seviteronel in subjects with castration-resistant prostate cancer (CRPC). Phase 1 was a dose-escalation study enrolling subjects with CRPC that were either "treatment naïve" (not treated with previous abiraterone or enzalutamide), or treated with one or more of the following: abiraterone, enzalutamide, or chemotherapy.

Phase 2 is an open-label, multi-center cohort-expansion study to further determine the efficacy and safety of seviteronel in two CRPC populations with documented rising PSA with or without bone or soft tissue disease progression during treatment with: abiraterone or enzalutamide for ≥ 12 weeks (Group 1) abiraterone and enzalutamide; treatment should be ≥ 12 weeks for at least one agent (Group 2)

ELIGIBILITY:
Inclusion Criteria:

1.18 years of age or older 2. Able to provide written informed consent or have their legal representatives provide written informed consent 3. Documented histological or cytological evidence of adenocarcinoma of the prostate. Subjects whose pathology reports are no longer available may be enrolled if, in the opinion of the investigator, the subject has a clinical course consistent with prostatic adenocarcinoma 4. ECOG Performance Status of 0 or 1 5. Undergone orchiectomy, or have ongoing LHRH analogue therapy prior to C1D1. Subjects on LHRH analogues should remain on these agents for the duration of the study 6. Castrate levels of testosterone less than or equal to 50 ng/dl (or 1.7 nmol/L) and have progressive disease at Screening defined as PSA rise determined by a minimum of 2 rising PSA values greater than or equal to 1 week between each assessment. The PSA value at the Screening visit must be greater than or equal 2ng/mL with or without: Soft tissue disease progression defined by RECIST 1.1 at Screening or less than or equal to 28 days of C1D1. Measurable disease is not required for entry.

Lymph nodes greater than or equal to 1.5cm (short axis) are considered measurable disease bone disease progression defined by greater than or equal 2 new lesions on bone scan at Screening, or less than or equal 28 days of C1D1 7. Have received abiraterone and/or enzalutamide. Subject must have received either abiraterone or enzalutamide for greater than or equal to 12 weeks. Other second generation CYP17 inhibitors/androgen receptor antagonists including but not limited to TAK-700 (orteronel), TOK-001 (galeterone) may have been taken in place of abiraterone and ARN-509 (apalutamide) may have been taken in place of enzalutamide.

8. Adequate hematopoietic function as evidenced by:

* WBC greater than or equal to 3,000/μl
* ANC greater than or equal to 1,500/μl
* Platelet count greater than or equal to 100,000/μl
* HGB greater than or equal to 10 g/dl and not transfusion dependent 9. Adequate liver function, including all the following:
* Total serum bilirubin less than or equal to 2.0 x ULN unless the subject has documented Gilbert syndrome;
* Aspartate and alanine aminotransferase (AST & ALT) less than or equal to 3.0 x ULN or less than or equal to 5.0 x ULN if subject has liver metastasis;
* Alkaline phosphatase less than or equal to 3.0 x ULN or less than or equal to 5 x ULN in case of bone metastasis and/or hepatic metastasis 10. Subjects must have adequate renal function as evidenced by a serum creatinine of less than or equal to 2.0 mg/dl 11. Potassium (K+) greater than or equal to 3.5 mEq/l 12. Subject and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at Screening and continuing throughout the study period and for 3 months after final study drug administration.
* Two acceptable forms of birth control include:

  1. Condom (barrier method of contraception), and
  2. One of the following:

     1. Oral, injected or implanted hormonal contraception
     2. Placement of an intrauterine device (IUD) or intrauterine system (ISU)
     3. Additional barrier methods of contraception: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
     4. Vasectomy or surgical castration greater than or equal to 6 months prior to Screening.

  13. Able to swallow study medication 14. Able to comply with study requirements

Exclusion Criteria

Each subject eligible to participate in this study must not have any of the following:

1. Received sipuleucel-T (Provenge ®) treatment within 28 days of C1D1
2. Received 5-alpha reductase inhibitors such as finasteride (PROSCAR®, PROPECIA®), or dutasteride (AVODART®) within 28 days of C1D1
3. Received any investigational agent less than or equal to 28 days of C1D1
4. Received palliative radiotherapy less than or equal to 2 weeks of C1D1
5. Symptomatic CNS metastases
6. History of another invasive malignancy less than or equal to 3 years of C1D1
7. A QTcF interval of greater than 470 msec; if the Screening ECG QTcF interval is greater than 470 msec, it may be repeated, and if repeat less than or equal to 470 msec, the subject may be enrolled
8. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes, second degree or third degree atrioventricular heart block without a permanent pacemaker in place)
9. Started a bone modifying agent (e.g. bisphosphonates, denosumab) less than or equal to 28 days of C1D1 (note: ongoing bone modifying agents administered less than 28 days are allowed)
10. Any medical condition that could preclude subject participation in the study, pose an undue medical hazard, or which could interfere with study results
11. Class III or IV Congestive Heart Failure (CHF) as defined by the New York Heart Association (NYHA) functional classification system within the previous 6 months
12. A history of loss of consciousness or transient ischemic attack less than or equal to 12 months of C1D1
13. Known active HIV, Hepatitis B, or Hepatitis C infections
14. Known or suspected hypersensitivity to seviteronel, or any components of the formulation
15. Any other condition which in the opinion of the investigator would preclude participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2011-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have ≥50% PSA decline at any time on study from the start of treatment with seviteronel. | 6 months
  Review of subjects with defined PSA value decline of greater than or equal to 50% from study start.
Median time to radiographic disease progression evaluated by computerized tomography (CT scan) or magnetic resonance imaging (MRI) and radionuclide bone scans by RECIST 1.1 | 10 months
  Review of subject disease progression status via CT and measure of median time to progression if progression occurs.

SECONDARY OUTCOMES:
Radiographic response rate by RECIST 1.1 & PCWG3. Safety of seviteronel with or without concurrent glucocorticoid administration | 10 months
  Evaluate RECIST 1.1 response and PCWG3 guidelines for responses.

OTHER OUTCOMES:
Determine biomarkers for response to seviteronel (e.g., circulating tumor DNA (ctDNA) for AR-v7) | 10 months
  Determine if biomarkers are predictors of response to study treatment

CONTACTS AND LOCATIONS:
Locations (23):
- United States (19):
  - Urology Centers of Alabama, Homewood, Alabama
  - H. Lee Moffitt Cancer and Research Institute, Tampa, Florida
  - First Urology, PSC, Jeffersonville, Indiana
  - Wichita Urology, Wichita, Kansas
  - Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - NY Cancer and Blood Specialists, The Bronx, New York
  - Duke Cancer Institute at Cary: Medical Oncology, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Alexandria Hospital, Department of Oncology, Athens, Greece
- Kantonsspital St Gallen, Onkologie/ Hamatologie, Sankt Gallen, Canton of St. Gallen, Switzerland
- United Kingdom (2):
  - The Royal Marsden Hospital - Institute of Cancer Research, Sutton, Surrey
  - Guys and St. Thomas' NHS Foundation Trust, London